CLINICAL TRIAL: NCT07086885
Title: Strength Training Intervention for Hybrid Workers: A Randomised Pilot Feasibility Trial
Brief Title: Strength Training Intervention for Hybrid Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Gemma Ryde, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200210134
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Strength; Productivity; Stress; Work Engagement
Keywords: Workplace; health promotion; resistance training; stress; productivity; work engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual routine
- Resistance band training (Experimental)
  Interventions: Behavioral: Resistance band training

INTERVENTIONS:
Behavioral: Resistance band training — Four-week resistance band training intervention (15 mins 3x per week). Written and video instructions on the exercises were provided inlcuding guidance on increasing resistance over the weeks.
  Arms: Resistance band training

SUMMARY:
What Is This Study About? To find out if a short, easy-to-do resistance band workout can help people who work both at home and in the office feel stronger, less stressed, and more productive.

What Can Be learnt?

* Can doing resistance band exercises make people physically stronger?
* Can it help reduce stress and improve how well people work? How Will the Study Work?

Two groups will be compared:

* One group will do resistance band exercises.
* The other group won't change anything in their routine. What Will Participants Do?
* A 15-minute resistance band workout three times a week for four weeks
* Complete a short strength test and survey before and after the 4 weeks
* Send in a weekly training diary by email

ELIGIBILITY:
Inclusion Criteria:

* working from home in the United Kingdom
* working from home 3 or more days per week
* performing less than 2 days per week of muscle strengthening exercise

Exclusion Criteria:

* Not working from home
* Working outside the United Kingdom
* performing more than 2 days per week of muscle strengthening exercise
* on holiday during the study
* answered yes to any of the questions in the Physical Activity Readiness Questionnaire

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Sit to stand | at baselines and then one week after the intervention ended
  Number of sit to stands in 30 seconds - Higher score are positive
Push-up | Baseline and one week after the intervention
  Number of push ups in 30 seconds - Higher scores are positive

SECONDARY OUTCOMES:
Stress | Baselines until one week after the intervention
  Perceived stress was measured using the 10 item Cohen-Perceived Stress Scale. This instrument is designed to measure psychological stress and to evaluate the stressful situations of daily life by measuring the degree an individual feels their life has been unpredictable, uncontrollable and overloaded during the past month. Questions were rated on a five-point Likert scale ranging from never (0) to almost always (4) with the ratings for each question summed to create an overall stress score. Higher scores indicate more perceived stress with the possible range of summed scores ranging from zero to 40. Scores of 13 are classified as average stress levels and scores of 20 or above indicate high stress levels.
Productivity | Baselines until one week after the intervention
  The Health and Work Questionnaire (HWQ) measures employee productivity and health. The survey consists of 24 questions (3 with sub-questions) used to create an overall HWQ score and six subscales; productivity, concentration/focus, supervisor relations, impatience/irritability, work satisfaction, and non-work satisfaction. Questions are rated on a 10-point Likert scale from a negative rating (1) to a positive rating (10). Scores for each subscale are calculated from the sum of responses to all the items comprising the subscale divided by the number of items in the subscale. An overall HWQ score is produced from the average of all six subscales. Scores closer to 10 indicate desirable productivity outcomes.
Work engagement | Baselines until one week after the intervention
  The Utrecht Work Engagement Scale (UWES) measures work engagement, which can be described as the opposite of burnout. The UWES-17 consists of 17 statements used to create an overall engagement score and three subscales: vigor, absorption, and dedication. Statements are rated on a 7-point Likert scale from never had this feeling (0) to always every day (6). Scores for each subscale are calculated from the sum of responses to all the items within that subscale, divided by the number of items in the subscale. An overall engagement score is produced from the average of all 17 subscales. Normative scores range from very low to very high, with very low scores for vigor, dedication, absorption and total engagement reported as ≤2.17, ≤1.60, ≤1.60 and ≤1.93, respectively, and very high scores reported as ≥5.61, ≥5.80, ≥5.36 and ≥5.54, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Annonymised participant data will be made available by the author upon request.
Supporting Information: Study Protocol
Time Frame: Data and study protocol will be made available as part of publication.